CLINICAL TRIAL: NCT04397614
Title: Mobile Health Study and Enhanced Symptom Monitoring to Prevent Severe Illness From COVID-19 in Cancer Patients
Brief Title: Mobile Health Study and Enhanced Symptom Monitoring in COVID-19 Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: COVID-19 Mobile Health; 3P30CA225520-03S3 (NIH)
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Sars-CoV2; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Elevated Risk for COVID-19 Detected (Experimental): Continue daily mHealth assessments
  Interventions: Other: mHealth Assessments
- Elevated Risk for COVID-19 Detected (Experimental): Daily mHealth assessments and telemedicine/nurse triage. If non-emergent intervention, enhanced symptom monitoring will occur.
  Interventions: Other: mHealth Assessments

INTERVENTIONS:
Other: mHealth Assessments — Daily symptom tracker

SUMMARY:
The established Insight(TM) mHealth Platform, a component of the Stephenson Cancer Center (SCC) mHealth Shared Resource will be used to create the "Symptom Tracker" app. The Symptom Tracker (Insight(TM)) app will enable real-time monitoring of cancer patient symptoms that are consistent with early signs of SARS-CoV-2 infection in this high-risk population by automatically (and securely) transferring this information to health care providers. The primary aim of this study is to determine the feasibility, ease of use, and perceived utility of this app to monitor symptoms and health risk behaviors among cancer patients currently receiving chemotherapy.

DETAILED DESCRIPTION:
A total of 500 treatment-seeking males and females will be asked to complete daily monitoring of symptoms via smartphone app. Those who screen positive for COVID-19 will be triaged to emergency or non-emergency medical treatment and will receive a study supplied device to measure their oxygen level and heart rate and be instructed in the device's use. They will be prompted to enter vital signs data (such as oxygen level) daily (and as indicated by changes in status) and questions from the app will change to assess the severity of COVID-19 related symptoms and inform changes in level of care, to emergency or non-emergency medical management as indicated by self-reporting. The proposed study will assess the impact of heightened symptom and vital sign monitoring on the early identification of severe manifestations of COVID-19 in this high-risk population (Aim 2). It is hypothesized that this will significantly improve COVID-19 related morbidity and mortality compared to the national and international rates currently reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrate > 6th grade English literacy level (i.e., phone based EMAs require >6th grade literacy)
2. Present for care at the Stephenson Cancer Center at the University of Oklahoma Health Sciences Center
3. Are currently receiving systemic chemotherapy by intravenous infusion or by orally delivered medication
4. Are greater than or equal to 18 years of age
5. Are willing and able to complete surveys on their personal smartphone or a study provided smartphone
6. Are willing and able to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Hannafon, PhD, Principal Investigator — The University of Oklahoma Health Sciences Center; Michael Businelle, PhD, Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Started | 121 | 7
Completed | 57 | 4
Not Completed | 64 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected | Total
Number analyzed (Participants) | 121 | 7 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.56) | 50.71 (12.56) | 57.60 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 5 | 99
  Male | 27 | 2 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 2 | 11
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 1 | 9
  White | 95 | 4 | 99
  More than one race | 7 | 0 | 7
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Smartphone Based Surveys Completed
Description: Proportion of completed smartphone-based daily surveys divided by the total number of surveys a participant is staged to receive (daily for 24 weeks = 168 surveys total)
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: proportion of daily surveys completed
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 121 | 7
proportion of daily surveys completed | 0.46 (0.38) | 0.44 (0.25)

2. Primary Outcome: Number of Participants With Manifestations of Severe Disease
Description: Yes/No; Yes = there were manifestations of severe disease; No = there were no manifestations of severe disease. Those who are marked as Yes are reported below in the Outcome measure data table
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 121 | 7
Participants | 25 | 5

3. Primary Outcome: Number of Participants With SARS-CoV-2 Related Hospital Admission
Description: Yes/No; Yes = there were SARS-CoV-2 related hospital admissions; No = there were no SARS-CoV-2 related hospital admissions. Those who are marked as Yes are reported below in the Outcome measure data table
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 121 | 7
Participants | 5 | 1

4. Primary Outcome: Number of Participants With SARS-CoV-2 Related ICU Admission
Description: Yes/No; Yes = there were SARS-CoV-2 related ICU admissions; No = there were no SARS-CoV-2 related ICU admissions. Those who are marked as Yes are reported below in the Outcome measure data table
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 121 | 7
Participants | 0 | 1

5. Primary Outcome: Number of Participants With SARS-CoV-2 That Needed Invasive Mechanical Ventilation
Description: Yes/No; Yes = participant had SARS-CoV-2 and needed invasive mechanical ventilation; No = participant had SARS-CoV-2 and did not need invasive mechanical ventilation. Those who are marked as Yes are reported below in the Outcome measure data table
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 121 | 7
Participants | 0 | 0

6. Primary Outcome: Mortality Number for Participants Who Reported SARS-CoV-2 Positive and Got Enhanced Monitoring
Description: Yes/No; Yes = participant mortality reported; No = participant mortality not reported. Those who are marked as Yes are reported below in the Outcome measure data table
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 121 | 7
Participants | 6 | 1

7. Secondary Outcome: Percent of Participants Satisfied With Monitoring and Use of mHealth Application
Description: 1. if the participants were satisfied with the number of assessments prompted by the smartphone application - yes/no - those who reported yes are in the outcome measure data table below
  2. if the participants would be interested in using a similar smartphone app in the future if needed - yes/no - those who reported yes are in the outcome measure data table below
Time Frame: 24 weeks
Population: Participants who completed the follow-up assessments
Measure: Count of Participants; unit: Participants
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
Number analyzed (Participants) | 57 | 4
Participants
  satisfied with number of assessments | 49 | 3
  interested in using a similar smartphone app if needed | 47 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the duration of the study for each participant, up to 24 weeks.
Arm/Group | No Elevated Risk for COVID-19 Detected | Elevated Risk for COVID-19 Detected
All-Cause Mortality (participants affected / at risk) | 6/121 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/7
Other Adverse Events (participants affected / at risk) | 0/121 | 0/7

LIMITATIONS AND CAVEATS:
None to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT04397614/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT04397614/ICF_001.pdf